CLINICAL TRIAL: NCT01795508
Title: The Effect of Parent Management Training, Oregon, in Denmark
Brief Title: Parent Management Training, Oregon
Acronym: PMTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIVE - The Danish Center for Social Science Research (Other)
Collaborators: National Board of Social Services, Denmark (Unknown); Ministry of Social Affairs, Denmark (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFI 2505
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Child Behavior Problems
Keywords: Parent training; Child behavior; Randomized Controlled Trials
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PMTO (Experimental): Parent Management Training Oregon
  Interventions: Behavioral: PMTO
- TAU (Active Comparator): Other kinds of family treatment
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: PMTO — Parent Management Training, Oregon
  Arms: PMTO
Behavioral: TAU — Other kinds of family training
  Arms: TAU

SUMMARY:
The purpose of the study is to examine the effects of Parent Management Training Oregon (PMTO) compared to treatment as usual (TAU) for parents with children aged 3 and 12 showing behavioral problems.

DETAILED DESCRIPTION:
This project estimates the causal effect of Parent Management Training, Oregon (PMTO) in a Danish context. The study design is an RCT where PMTO is compared to Treatment As Usual (TAU). The target population is parents with children aged 3 and 12 showing behavioral problems. The primary outcome estimates changes in child behavior, and is measured three times: baseline, seven months follow-up, and 19 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Families with children that are eligible for PMTO and at least one other type of family training program

Exclusion Criteria:

* The family does not want to participate

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Strength and Difficulties Questionnaire (SDQ) | 7 months post baseline
  Measuring child behavior
Brief Problem Monitor-Parent Form (BPM-P) | 7 months post baseline
  Measuring child behavior

SECONDARY OUTCOMES:
Parents Preference Test (PPT) | 7 months post baseline
  Parenting skills
Sense of Coherence (SOC) | 7 months post baseline
Parental Stress Scale (PSS) | 7 months post baseline
Parenting Sense of Competence scale (PSOC) | 7 months post baseline
Major Depression Inventory (MDI) | 7 months post baseline

CONTACTS AND LOCATIONS:
Locations (1):
- SFI the Danish National Centre for Social Research, Copenhagen, Copenhagen K, Denmark